CLINICAL TRIAL: NCT01238094
Title: Placebo-controlled, Double-blinded Phase III Trial of XELIRI/FOLFIRI + Simvastatin Followed by Simvastatin Maintenance in Metastatic Colorectal Cancer
Brief Title: Trial of XELIRI/FOLFIRI + Simvastatin Followed by Simvastatin Maintenance in Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009-11-017
Record Dates: First submitted 2010-06-22; First posted 2010-11-10 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2012-01

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; simvastatin; second-line chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFIRI or XELIRI/simvastatin (Experimental): FOLFIRI or XELIRI/simvastatin
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — simvastatin 40 mg qd daily until disease progression

SUMMARY:
The purpose of this study is to compare 2nd line XELIRI/FOLFIRI + simvastatin vs XELIRI/FOLFIRI + placebo.

DETAILED DESCRIPTION:
To compare progression free survival of the standard second line chemotherapy (FOLFIRI, XELIRI) plus simvastatin in metastatic colorectal cancer patients. This trial is a placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented colorectal adenocarcinoma (previously failed to oxaliplatin)
2. Age over 19 years old
3. Performance status (ECOG scale): 0-2
4. Measurable or evaluable disease
5. Adequate organ functions
6. Life expectancy ≥ 3 months
7. No history of statin treatment within the last 12 months
8. Patients should sign a written informed consent before study entry.

Exclusion Criteria:

1. Tumor type other than adenocarcinoma
2. Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin, papillary thyroid carcinoma or prior malignancy treated more than 5 years ago without recurrence)
3. Adjuvant or neo-adjuvant treatment for non-metastatic (M0) disease is allowed if completed at least 6 months prior to initiation of study treatment.
4. Prior radiotherapy is permitted if it was not administered to target lesions selected for this study, unless progression of the selected target lesions within the radiation portal is documented, and provided it has been completed at least 4 weeks before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-11 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Won Ki Kang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea